CLINICAL TRIAL: NCT04103008
Title: Effect of Residual Myocardial Ischemia on Recovery of Left Ventricular Function After Primary Percutaneous Coronary Intervention
Brief Title: Left Ventricular Function After Primary Percutaneous Coronary Intervention: Role of Speckle Echocardiography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karim Mohamed Eltaher Abdelrahman Aly, Resident of Cardiology, Assiut University
Other Study IDs: AssiutU2019
Record Dates: First submitted 2019-09-21; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Myocardial Infarction; Echocardiography 2D; Left Ventricular Dysfunction
Keywords: Speckle tracking; 2D echocardiography; Left ventricle residual function; PCI, percutaneous coronary intervention; single coronary artery; multiple coronary arteries
MeSH Terms: conditions — Myocardial Infarction; Ventricular Dysfunction, Left | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: single coronary artery lesion
  Interventions: Diagnostic Test: Speckle tracking echocardiography
- Group B: multiple coronary artery lesions
  Interventions: Diagnostic Test: Speckle tracking echocardiography

INTERVENTIONS:
Diagnostic Test: Speckle tracking echocardiography — assess left ventricular function on admission and after 40 days
  Other Names: 2 D echocardiography

SUMMARY:
Recovery of the left ventricular function is variable from one patient to another, thus assessment of cardiac function by measuring left ventricular ejection fraction using echocardiography is the most common in the daily clinical practice. However, this technique has limitation related with its intra- and interobserver variability. A recent technique, 2D speckle tracking for assessing global longitudinal strain, has been introduced to reduce the variability and potentially has a higher accuracy. Speckle tracking is a method which uses two dimensions recording for measuring quantity of movement of myocardium in several segments.

Speckle-tracking echocardiography is a current noninvasive ultrasound imaging technique that allows for an objective and quantitative evaluation of global and regional myocardial function independently from the angle of insonation and from cardiac translational movements,

DETAILED DESCRIPTION:
Authors using 2D speckle tracking found that subclinical LV systolic dysfunction is common in patients with isolated severe mitral stenosis (MS) and is determined primarily by the hemodynamic variables of MS severity and reduced LV filling. BMV results in rapid recovery of LV systolic function in these patients through improvement in LV diastolic loading. These findings suggest that LV contractile properties in MS are modulated predominantly by LV diastolic filling rather than myocardial structural abnormality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myocardial infarction eligible for PCI seen on admission and after 40 days

Exclusion Criteria:

* cardiomyopathy
* cancer
* on cytostatic treatment.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction with single or multiple coronary artery lesions seen after PCI on admission and after 40 days
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessing change of left ventricular function | baseline and after 40 days of PCI
  measure ejection fraction

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 40 days
  non fatal myocardial infarction, non fatal stroke, CV death

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Youssef, MD, Study Chair — Professor of Cardiology; Mohamed A Abdel Hafez, MD, Study Director — Associate Professor
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdelhafez MA, Aly KME, Youssef AAA. Effect of residual myocardial ischemia on recovery of left ventricular function after primary percutaneous coronary intervention. BMC Cardiovasc Disord. 2024 Mar 19;24(1):164. doi: 10.1186/s12872-024-03777-3. PMID 38504186